CLINICAL TRIAL: NCT06978868
Title: The Effect of Sauna on Cardiac and Skeletal Muscle Function in Patients With HFpEF (SAUNA-HFpEF): A Mechanistic, Pilot Prospective, Single-arm, Single Centre Study
Brief Title: Effects of Sauna on Cardiac and Skeletal Muscle Function in Patients With HFpEF (SAUNA-HFpEF)
Acronym: SAUNA-HFpEF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Otto-von-Guericke University Magdeburg (Other)
Responsible Party: Principal Investigator, Tarek Bekfani, Associate Professor Tarek Bekfani, MD, MSc (Oxon.), FESC, FHFA, Otto-von-Guericke University Magdeburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 61/23
Record Dates: First submitted 2025-04-17; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Heart Failure With Preserved Ejection Fraction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinically stable outpatients with HFpEF (Experimental): All participants will be accompanied by medical doctors for two sessions weekly, each between 8-15 minutes. The intervention will be done in the NEMO-sauna in Magdeburg. The duration of the intervention will be 10 weeks. We will start the first 2 weeks with 8 minutes. Week 3-4: 10 minutes, week 5-6: 12 minutes, week 7-10: 12-15 minutes. Sessions will be done in groups each consisting of 5 patients. The temperature of the sauna will be 60°C. After each session a cold shower will follow and then rest for 20 minutes. Blood pressure, heart frequency, O2-Saturation will be measured prior to each session as well as directly after the shower and at the end of the rest.
  Interventions: Other: Sauna Intervention in Clinically Stable Outpatients with HFpEF

INTERVENTIONS:
Other: Sauna Intervention in Clinically Stable Outpatients with HFpEF — Patients were accompanied by study physicians for two sessions weekly, each between 8-15 minutes. We started the first 2 weeks with 8 minutes. Week 3-4: 10 minutes, week 5-6: 12 minutes, week 7-10: 12-15 minutes. Patients were given the freedom to leave the sauna session at any time if they experienced discomfort or were unable to tolerate it. Sessions were done in groups of 5 patients of men or women. The temperature of the sauna was 60°C. After each session, patients were asked to shower with moderate temperature of water and then rest for 20 minutes. Blood pressure and heart rate were measured prior to each session as well as directly after the sauna session and at the end of the rest time.

SUMMARY:
Heart failure with preserved ejection fraction (HFpEF) is a type of heart failure where the heart pumps normally but patients still experience symptoms like fatigue, shortness of breath, and reduced ability to exercise. Many patients with HFpEF also have muscle weakness and limited mobility, which makes it difficult to follow traditional exercise programs like running or cycling. While there have been improvements in treating other types of heart failure, finding effective options for this specific form remains a challenge.

This study will explore whether bio-sauna bathing-a form of mild heat therapy-can help improve muscle function and exercise ability in patients with HFpEF. Sauna therapy might offer similar benefits to light exercise and could be easier and safer for older patients or those who can't do intense physical activity. The goal of this study is to evaluate whether regular sauna sessions is safe in patients with HFpEF and if it can improve exercise capacity, reduce shortness of breath, and support muscle health in patients with HFpEF.

DETAILED DESCRIPTION:
The aim of the study is to test the safety and efficacy of intermittent hyperthermia (sauna) in a pilot study on patients with HfpEF regarding cardiac function, exercise capacity, skeletal muscle structure and function, metabolomic changes, and quality of life both at baseline and after the intervention with sauna.

Hypothesis: It was hypothesized that intermittent hyperthermia (sauna) is a feasible intervention in patients with HFpEF. Explorative, the effect of the intervention on filling pressure (E/é) as well as on the level of NT-pro-BNP, will be tested. Peripherally, skeletal muscle function (including metabolic and mitochondrial function) and structure. Finally, the effects of the intervention on QoL will be tested.

Questions to be answered through our investigation,

1. Is hyperthermia intervention (sauna) feasible in patients with HF?
2. Does sauna improve exercise capacity? (CPET, 6MWT, skeletal muscle strength and endurance).
3. Does sauna improve cardiac function (Echocardiography).
4. Understanding the related pathophysiology of the observed results on skeletal muscle and exercise capacity on molecular and mitochondrial level (skeletal muscle biopsies and the following tissue analysis parallel to blood analysis).
5. The role of inflammation in the altered muscle structure and function and its possible reversibility through sauna.
6. Observing changes in QoL and mental health (depression and anxiety).

The results of this study will be supportive in planning the randomised controlled clinical trial.

The intervention was twice weekly for a period of 10 weeks. : All participants will undergo a standardized series of assessments such as echocardiogram, CPET, 6-MWT, muscle strength measurements, and skeletal muscle biopsies. In case of clinical improvement, these benefits are likely to diminish over time if sauna bathing is discontinued. To address this, patients will be invited for a follow-up visit three months after completing the intervention. All investigations will be repeated, except for the skeletal muscle biopsy.

ELIGIBILITY:
Inclusion criteria:

* NYHA class II or III, clinically stable in the previous three months
* Females and males, age >50 years
* Left ventricular EF >50%, and at least 2 of the following: left atrial volume index (LAVI ≥34ml/m2) or E/e' >9 or interventricular septal thickness >12mm or pulmonary arterial pressure >35mmHg (noninvasive measurement) for HFpEF as recommended according to the ESC-HF-guidelines.
* Stable on standard HF medication according to the ESC-HF guidelines in the last 4 weeks

Exclusion criteria:

* Major cardiovascular event or procedure such as myocardial infarction, percutaneous coronary intervention (PCI), aortocoronary bypass operation in the previous 3 months.
* Patients who have an indication for dual platelet inhibition
* Stroke
* Patients with mechanical heart valves or implanted cardiac devices
* Pulmonary embolism or deep vein thrombosis
* Patients with altered or reduced sweat function, such as in autoimmune diseases, spinal cord injuries or Fabry disease
* Symptomatic hypotension regardless of the measured value and those with BP systolic <110 mm Hg
* Patients on oral anticoagulation for other reasons than atrial fibrillation
* Uncontrolled diabetes mellitus (HbA1c>8%), severe renal dysfunction, GFR<30ml/min) or pulmonary disease (COPD GOLD ≥3)
* Primary muscle disorder (e.g., muscular dystrophies)
* Neurological disease (e.g., Dementia or Parkinson syndrome)
* Right ventricular dysfunction or uncontrolled arrhythmias
* Any condition that in the opinion of the investigator could prohibit performance of 6MWT

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-10-19 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-08-16 (Actual)

PRIMARY OUTCOMES:
Exercise capacity | 10 weeks
  The clinical effect of sauna on peak VO2 (ml/min)

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Bekfani, MD, MSc, Principal Investigator — University Hospital Magdeburg
Locations (1):
- Otto von Guericke University, Faculty of Medicine, Magdeburg, Saxony-Anhalt, Germany

DOCUMENTS (1):
  • Study Protocol (2024-06-06): https://cdn.clinicaltrials.gov/large-docs/68/NCT06978868/Prot_000.pdf